CLINICAL TRIAL: NCT07350226
Title: Efficacy and Amygdala-entorhinal Circuit of Electroacupuncture Intervention in SCD With Depression: A Randomized Controlled Trial
Brief Title: Electro-acupuncture for SCD With Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JSTJ-2024-381
Record Dates: First submitted 2025-12-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Subjective Cognitive Decline (SCD); Depression Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): "TXJN" electro-acupuncture：Disposable acupuncture needles (Huatuo brand, Suzhou Medical Supplies Factory Co., Ltd., specification: 0.25 mm × 40 mm) were used.The selected acupoints included bilateral Neiguan (PC6), Yintang (EX-HN3), bilateral Yingxiang (LI20), Shenting (GV24), Baihui (GV20), and Sishencong (EX-HN1).After achieving the deqi sensation through acupuncture manipulation, electroacupuncture (SDZ-V, Huatuo brand, Suzhou Medical Supplies Factory Co., Ltd.) was applied. The treatment utilized a dense-disperse wave at a frequency of 2 Hz, with a current intensity of 2-4 mA adjusted to the patient's tolerance level. The needles were retained for 30 minutes.The treatment was administered once daily, 3-5 times per week, for a total duration of 8 weeks.
  Interventions: Device: "TXJN" electro-acupuncture
- Control group (Sham Comparator): Sham electroacupuncture: Disposable acupuncture needles (Huatuo brand, Suzhou Medical Supplies Factory Co., Ltd., specification: 0.25 mm × 40 mm) were used.Acupoints were selected at 0.2-0.4 cun (5-10 mm) lateral to the original acupoints of the experimental group. The needles were inserted shallowly at a depth of 0.2-0.3 cun (5-8 mm), without eliciting the deqi sensation. The same electroacupuncture device was connected but with no electrical output. The needles were retained for 30 minutes.The treatment was administered once daily, 3-5 times per week, for a total duration of 8 weeks.
  Interventions: Device: Sham electroacupuncture

INTERVENTIONS:
Device: "TXJN" electro-acupuncture — Disposable acupuncture needles (Huatuo brand, Suzhou Medical Supplies Factory Co., Ltd., specification: 0.25 mm × 40 mm) were used.
  The selected acupoints included bilateral Neiguan (PC6), Yintang (EX-HN3), bilateral Yingxiang (LI20), Shenting (GV24), Baihui (GV20), and Sishencong (EX-HN1).After achieving the deqi sensation through acupuncture manipulation, electroacupuncture (SDZ-V, Huatuo brand, Suzhou Medical Supplies Factory Co., Ltd.) was applied. The treatment utilized a dense-disperse wave at a frequency of 2 Hz, with a current intensity of 2-4 mA adjusted to the patient's tolerance level. The needles were retained for 30 minutes.The treatment was administered once daily, 3-5 times per week, for a total duration of 8 weeks.
  Arms: Experiment group
Device: Sham electroacupuncture — Disposable acupuncture needles (Huatuo brand, Suzhou Medical Supplies Factory Co., Ltd., specification: 0.25 mm × 40 mm) were used.Acupoints were selected at 0.2-0.4 cun (5-10 mm) lateral to the original acupoints of the experimental group. The needles were inserted shallowly at a depth of 0.2-0.3 cun (5-8 mm), without eliciting the deqi sensation. The same electroacupuncture device was connected but with no electrical output. The needles were retained for 30 minutes.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of electroacupuncture in treating adults with subjective cognitive decline accompanied by depression. The main objectives are to answer the following questions:

1. Can electroacupuncture improve cognitive function and depressive symptoms in individuals with subjective cognitive decline accompanied by depression?
2. Does electroacupuncture alleviate subjective cognitive decline with depression by modulating the amygdala-entorhinal circuit, and if so, what is the specific mechanism involved? Researchers will compare real electroacupuncture therapy with sham electroacupuncture therapy to determine whether real electroacupuncture can effectively improve symptoms in patients with subjective cognitive decline accompanied by depression. Additionally, multimodal magnetic resonance imaging (MRI) technology will be used to assess changes in the amygdala-entorhinal circuit following electroacupuncture intervention.

Participants will:

1. Receive either real or sham electroacupuncture treatment once daily, 3-5 times per week, for a total treatment duration of 8 weeks.
2. Undergo cognitive function and depression assessments before and after treatment.
3. Complete multimodal cranial magnetic resonance imaging examinations before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80 years, right-handed
* Meets the diagnostic criteria for Subjective Cognitive Decline (SCD)
* Geriatric Depression Scale-15 (GDS-15) score ≥5
* Clear consciousness, cooperative during examination, with adequate auditory comprehension
* Patient and family agree to complete assessments and have provided informed consent with signed documentation

Exclusion Criteria:

* Received other anti-dementia or antidepressant therapy within the past 2 weeks, or currently participating in other clinical trials
* Experienced acute cerebral infarction, cerebral hemorrhage, or transient ischemic symptoms within the past 6 months, or presence of localized old encephalomalacia foci
* History of positive neuropsychiatric disorders and major trauma, including dementia, depression, epilepsy, etc.
* Suffering from other severe comorbidities (aphasia, diabetic ketoacidosis, hyperosmolar hyperglycemic state, diabetic lower limb vascular disease, moderate to severe edema of lower limbs, lower limb venous thrombosis, arteriosclerosis obliterans of lower limbs, peripheral neuropathy, spinal cord lesions, traumatic brain injury, intracranial infection, brain tumors, etc.) or secondary diseases (e.g., heart, liver, or renal failure, etc.)
* Infection at the acupuncture site and/or intolerance to acupuncture therapy
* Contraindications to MRI examination (claustrophobia, surgically implanted metal devices, cochlear implants, implanted pulse generators, etc.)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Cognitive Z-Score | Before and 8 weeks after treatment
  This composite index of global cognitive function is derived from the aggregated Z-scores of eight neuropsychological tests (including Auditory Verbal Learning Test, Animal Fluency Test, Boston Naming Test, Trail Making Test Parts A/B, Stroop Color-Word Test-Card C, Digit Symbol Substitution Test, Digit Span Test, and Clock Drawing Test). At baseline, each test's raw scores will be standardized using the study population's mean and standard deviation (Z = [raw score - mean]/SD). For tests where lower scores indicate better performance (e.g., Trail Making Test time), Z-scores are reversed (multiplied by -1) to align directionality. The final aggregated Z-score, expressed in standard deviation units, will be assessed pre-treatment and 8 weeks post-treatment initiation.
Geriatric Depression Scale 15-Item (GDS-15) Reduction Rate | Before and 8 weeks after treatment
  The reduction rate is calculated based on the total score (range: 0-15, where a higher score indicates more severe depressive symptoms) of the 15-item Geriatric Depression Scale. The reduction rate formula is: ([Pre-treatment score - Post-treatment score] / Pre-treatment score) × 100%. Efficacy is defined as: Markedly Effective (reduction rate ≥ 50%); Effective (50% > reduction rate ≥ 25%); Ineffective (reduction rate < 25%).
Multimodal magnetic resonance imaging indicators | Before and 8 weeks after treatment
  sMRI indicators: GMV, FA, MD; rs-fMRI indicators: ALFF, fALFF, ReHo, Seed-based FC.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) Total Score | Before and 8 weeks after treatment
  The total score (range: 0-30) of the Mini-Mental State Examination, where a higher score indicates better cognitive function.
Auditory Verbal Learning Test (AVLT) Long-Delay Free Recall Score | Before and 8 weeks after treatment
  The score for the long-delay free recall trial of the Auditory Verbal Learning Test (range: 0-15 words), where a higher score indicates better episodic memory function.
Rey-Osterrieth Complex Figure Test (ROCF) Delayed Recall Score | Before and 8 weeks after treatment
  The score for the delayed recall trial of the Rey-Osterrieth Complex Figure Test, which is typically scored on a standardized system (e.g., 0-36 points based on accuracy and placement of reproduced elements), where a higher score indicates better visual-spatial memory and recall ability.
Boston Naming Test (BNT) Total Correct Score | Before and 8 weeks after treatment
  The total number of correctly named items (range: 0-30) of the 30-item Boston Naming Test, where a higher score indicates better confrontational word retrieval and language ability.
Animal Fluency Test (AFT) Total Score | Before and 8 weeks after treatment
  The total number of correct, unique animal names generated within 60 seconds (common score range: 0-50+), where a higher score indicates better semantic verbal fluency and executive functioning.
Trail Making Test Part A (TMT-A) Completion Time | Before and 8 weeks after treatment
  The time to completion (in seconds) for Trail Making Test Part A, where a shorter completion time indicates better visual attention, processing speed, and motor function.
Trail Making Test Part B (TMT-B) Completion Time | Before and 8 weeks after treatment
  The time to completion (in seconds) for Trail Making Test Part B, where a shorter completion time indicates better cognitive flexibility, task-switching ability, and executive function.
Clock Drawing Test (CDT) Total Score | Before and 8 weeks after treatment
  The total score on the standardized 30-point Clock Drawing Test (CDT30-AJ/CI version, range: 0-30), where a higher score indicates better visuospatial/executive function and cognitive integrity.
Symbol Digit Modalities Test (SDMT) Correct Response Count | Before and 8 weeks after treatment
  The total number of correct symbol-digit pairings completed within 90 seconds (common score range: 0-110+), where a higher score indicates better processing speed, sustained attention, and visual scanning.
Pittsburgh Sleep Quality Index (PSQI) Global Score | Before and 8 weeks after treatment
  The global score (range: 0-21) of the Pittsburgh Sleep Quality Index, where a higher score indicates poorer sleep quality.
TCM Constitution Classification and Determination Scale - Transformed Scores | Before and 8 weeks after treatment
  The transformed scores (range: 0-100 for each of the nine constitution subscales) calculated according to the standardized "TCM Constitution Classification and Determination Scale" (published by the China Association of Chinese Medicine). A higher transformed score on a specific subscale indicates a more pronounced tendency towards that constitution type (e.g., Yang Deficiency, Qi Deficiency, etc.).
TCM Syndrome Type Scale for Mild Cognitive Impairment Subscale Scores | Before and 8 weeks after treatment
  Scores (range: 0-30 per syndrome) for seven TCM syndrome types (e.g., Spleen-Kidney Deficiency) as assessed by the standardized "TCM Syndrome Type Scale for Mild Cognitive Impairment", where a higher score indicates more severe syndrome manifestation.

OTHER OUTCOMES:
Treatment Acceptance Survey Response | After 8 weeks of treatment
  The participant's response to a single-item Treatment Acceptance Survey at the end of the treatment period. Responses are categorized as: "Completely Acceptable", "Acceptable", or "Not Acceptable".
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From treatment initiation up to 8 weeks.
  The number and proportion of participants experiencing any treatment-emergent adverse event(s), classified by system organ class and severity (e.g., mild, moderate, severe), according to a standardized dictionary (e.g., MedDRA) and assessed for relationship to the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes